CLINICAL TRIAL: NCT02996994
Title: Predictors of Postoperative Pain in Urogynecologic Surgery
Brief Title: Predictors of Postoperative Pain
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 16-093
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Results first posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective chart review using TriHealth Electronic Privacy Identification Center (EPIC) and previously developed databases for TriHealth Institutional Review Board (IRB) approved research studies within the Division of Urogynecology and Reconstructive Pelvic Surgery to determine the predictors of postoperative pain specific to the urogynecologic patient population.

DETAILED DESCRIPTION:
Postoperative pain remains the most important consideration for both patients and surgeons. Therefore, there has been much attention brought toward investigating predictive factors of postoperative pain. A systematic review of 48 eligible studies with 23,037 patients showed preexisting pain, anxiety, age, and type of surgery are the four most significant predictive factors for the intensity of postoperative pain. However, this paper evaluated all types of surgical approaches. More recently, a prospective observational study showed that preoperative State Trait Anxiety Inventory (STAI) and Numerical Rating Scales (NRS) for anxiety and pain expectations are independent predictors of pain and morphine consumption following abdominal hysterectomy. To date, little is known about the predictive factors of postoperative pain in the urogynecologic patient population.

The purpose of this study is to determine the predictors of postoperative pain specific to the urogynecologic patient population. We aim to investigate the relationship between perioperative factors (such as demographics and medical history) and postoperative pain scores on postoperative day 1 with patients who have undergone urogynecologic surgery, specifically vaginal reconstruction for pelvic organ prolapse.

This information would not only fill a gap in knowledge, but would also allow us to counsel our patients more accurately in regards to postoperative expectations. Furthermore, if we find any positive correlation between modifiable perioperative factors and postoperative pain scores, we may be able to minimize these effects in future surgical cases.

ELIGIBILITY:
Inclusion Criteria:

* Participant in one of six research studies previously performed by the Division of Urogynecology and Pelvic Reconstructive Surgery (#13090, #13072, #12136, #12132, #10072, or #09001)
* Postoperative pain scoring data complete and available
* Vaginal reconstructive surgery as primary treatment
* General anesthesia

Exclusion Criteria:

* Incomplete or unavailable postoperative pain scoring
* Robotic sacrocolpopexy patients will be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants of previous TriHealth IRB-approved research studies within the Division of Urogynecology and Reconstructive Pelvic Surgery that incorporated assessment of postoperative pain as part of the data collection
Sampling Method: Non-Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2016-12; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ip HY, Abrishami A, Peng PW, Wong J, Chung F. Predictors of postoperative pain and analgesic consumption: a qualitative systematic review. Anesthesiology. 2009 Sep;111(3):657-77. doi: 10.1097/ALN.0b013e3181aae87a. PMID 19672167
- [Background] Aouad MT, Kanazi GE, Malek K, Tamim H, Zahreddine L, Kaddoum RN. Predictors of postoperative pain and analgesic requirements following abdominal hysterectomy: an observational study. J Anesth. 2016 Feb;30(1):72-9. doi: 10.1007/s00540-015-2090-0. Epub 2015 Oct 24. PMID 26499321
- [Derived] Shatkin-Margolis A, Crisp CC, Morrison C, Pauls RN. Predicting Pain Levels Following Vaginal Reconstructive Surgery: Who Is at Highest Risk? Female Pelvic Med Reconstr Surg. 2018 Mar/Apr;24(2):172-175. doi: 10.1097/SPV.0000000000000522. PMID 29474293

RESULTS

PARTICIPANT FLOW:
Groups:
- Reconstructive Surgery: Eligible trials enrolled subjects undergoing vaginal reconstructive surgery for pelvic organ prolapse from 2009 to 2015.
Period: Overall Study
Arm/Group | Reconstructive Surgery
Started | 364
Completed | 364
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Reconstructive Surgery
Number analyzed (Participants) | 364
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.44 (11.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 364
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 351
  African American | 9
  Asian | 2
  Other | 1
  Missing | 1
Region of Enrollment [Number; unit: participants]
  United States | 364

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Pain Score
Description: VAS is a validated 100 millimeter scale with no pain as 0 mm and worst pain as 100 mm. Subjects drew a vertical line on the scale corresponding to their pain level.
Time Frame: postoperative day 1 (POD1)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Reconstructive Surgery
Number analyzed (Participants) | 364
mm | 38.16 (24.89)

ADVERSE EVENTS:
Time Frame: From time of surgery to 12 weeks after surgery
Arm/Group | Reconstructive Surgery
All-Cause Mortality (participants affected / at risk) | 0/364
Serious Adverse Events (participants affected / at risk) | 0/364
Other Adverse Events (participants affected / at risk) | 0/364

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT02996994/Prot_SAP_000.pdf